CLINICAL TRIAL: NCT07258589
Title: Taste and Smell Training in Patients With Cancer Who Are Treated With Tyrosine Kinase Inhibitors: a Multicentre Randomized Intervention Trial
Brief Title: The TASTY-training Study
Acronym: TASTY-training
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University Medical Center Groningen (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: 20901
Record Dates: First submitted 2025-11-20; First posted 2025-12-02 (Actual); Last update posted 2025-12-02 (Actual); Status verified 2025-11

CONDITIONS: Patients Who Are Treated With Tyrosine Kinase Inhibitors
MeSH Terms: interventions — Taste; Olfactory Training

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Taste and smell training (Experimental): To examine the effect of at-home taste and smell training versus standard care on taste function and other outcome parameters, measurements will take place at baseline (before the training starts), and after 12 weeks. The intervention will take place at home.
  Interventions: Behavioral: Taste and smell training
- No intervention (No Intervention): Standard of care

INTERVENTIONS:
Behavioral: Taste and smell training — To examine the effect of at-home taste and smell training versus standard care on taste function and other outcome parameters, measurements will take place at baseline (before the training starts), and after 12 weeks. The intervention will take place at home. The control group will receive usual care. Questionnaires will be filled in online at home, while taste and smell tests and saliva collection will be conducted either at home or in the hospital during regular visits. Patients in both study arms are contacted by their dietitian every 3 weeks.
  Arms: Taste and smell training

SUMMARY:
A multicentre non-blinded randomised intervention trial with a parallel cluster design. The multicentre study will be performed at 12 hospitals in the Netherlands. A parallel cluster design per hospital was selected to prevent contact between participants in the same hospital who are randomised into different study arms. Such contact may result in bias as it may allow for patients in the control arm to be informed about elements of taste and smell training.

To examine the effect of at-home taste and smell training versus standard care on taste function and other outcome parameters, measurements will take place at baseline (before the training starts), and after 12 weeks. The intervention will take place at home. The control group will receive usual care. Questionnaires will be filled in online at home, while taste and smell tests and saliva collection will be conducted either at home or in the hospital during regular visits. Patients in both study arms are contacted by their dietitian every 3 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥18 and ≤70 years
* Intention of being treated with tyrosine kinase inhibitors for next 12 weeks.
* Experiencing taste alterations after starting treatment with tyrosine kinase inhibitors
* Consuming solid foods and drinks is possible
* ≤50% of recommended daily intake in kcal consisting of oral nutritional supplements
* Oral mucositis grade ≤2 (Common Terminology Criteria for Adverse Events, version 5.0)
* Ability to comply with all protocol-required actions
* Written informed consent

Exclusion Criteria:

* Pregnancy
* History of taste, smell, or saliva production dysfunction before treatment with tyrosine kinase inhibitors
* Previous or current radiotherapy of head and neck region
* Enteral feeding through tube or parenteral feeding
* Participation in another clinical trial aimed at preventing or treating taste and/or smell alterations
* Chronic (>1 month) high dose corticosteroids (>10 mg prednisone/day or equivalent)

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 90 (Estimated)
Dates: Start 2025-11-10 (Actual); Primary Completion 2028-07 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Taste function | 12 weeks
  Taste function measured with taste strips at baseline and after week 12 weeks of taste and smell training compared with standard care

SECONDARY OUTCOMES:
Smell function | 12 weeks
  Smell function measured with Sniffin' Sticks at baseline and after week 12 of taste and smell training compared to standard care
Food enjoyment | 12 weeks
  Food enjoyment, measured by the subsection of the Appetite, Hunger and Sensory Perception Questionnaire and the Food enjoyment and food liking: questions on food enjoyment and food liking on 9-point hedonic scale at baseline and after 12 weeks of taste and smell training compared with standard care
Quality of life | 12 weeks
  Quality of life: EORTC QLQ-C30
Taste and smell alterations | 12 weeks
  Taste and smell alterations: Chemotherapy-induced Taste Alteration Scale (ciTAS-NL)
Risk of malnutrition | 12 weeks
  Risk of malnutrition: Patient-Generated Subjective Global Assessment (PG-SGA)
Dry mouth feeling | 12 weeks
  Dry mouth feeling: Xerostomia Inventory (XI) and Regional Oral Dryness Inventory (RODI)
Saliva secretion | 12 weeks
  Saliva secretion
Body weight | 12 weeks
  Body weight

CONTACTS AND LOCATIONS:
Overall Officials: J. J.A. de Haan, MD, PhD, Principal Investigator — University Medical Center Groningen
Locations (11):
- Netherlands (11):
  - Amsterdam UMC, Amsterdam
  - Rijnstate Ziekenhuis, Arnhem
  - Van Weel-Bethesda Ziekenhuis, Dirksland
  - Ziekenhuisvoorzieningen Gelderse Vallei, Ede
  - University Medical Center Groningen, Groningen
  - Martini Ziekenhuis, Groningen
  - Radboud University medical Center, Nijmegen
  - Ikazia Ziekenhuis, Rotterdam
  - Ommelander Ziekenhuis Groningen, Scheemda
  - Maxima Medisch Centrum, Veldhoven
  - Isala Klinieken, Zwolle